CLINICAL TRIAL: NCT02224079
Title: Safety, Tolerability and Preliminary Pharmacokinetics of Single Rising Doses of 1 mg, 2.5 mg, 5 mg, 10 mg, 15 mg, 20 mg, 25 mg, 37.5 mg, 50 mg, 75 mg, 100 mg, 125 mg and 150 mg BIIB 722 CL (Calculated as 'Free Base') and HPβCD Given as Intravenous Infusion Over 30 Minutes to Young Healthy Male Subjects. A Single-centre, Single-blind, Placebo-controlled, Randomised Study.
Brief Title: Safety, Tolerability and Pharmacokinetics of Single Rising Doses of BIIB 722 CL and HPβCD in Young Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1180.3
Record Dates: First submitted 2014-08-21; First posted 2014-08-25 (Estimated); Last update posted 2014-08-25 (Estimated); Status verified 2014-08

CONDITIONS: Healthy

ARMS (2):
- BIIB 722 CL (Experimental)
  Interventions: Drug: BIIB 722 CL; Drug: Placebo
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BIIB 722 CL
  Arms: BIIB 722 CL
Drug: Placebo — Hydroxypropyl-beta-cyclodextrin (HPβCD)

SUMMARY:
Study to assess safety, tolerability and pharmacokinetics (PK) of single intravenous (i.v.) doses of BIIB 722 CL

ELIGIBILITY:
Inclusion Criteria:

* Healthy males
* 21 to 50 years of age
* Broca index >= -20% and <= +20%
* Written informed consent according to Good Clinical Practice (GCP) and local legislation

Exclusion Criteria:

* Any finding of the medical examination (including blood pressure, pulse rate and Electrocardiogram (ECG)) deviating from normal and of clinical relevance
* History or current gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunologic or hormonal disorders
* Diseases of the central nervous system or psychiatric disorders or neurological disorders
* History of orthostatic hypotension, fainting spells or blackouts
* Chronic or relevant acute infections
* History of allergy/hypersensitivity (including drug allergy) which is deemed relevant to the trial as judged by the investigator
* Intake of drugs with a long half-life (> 24 hours) within at least one month or less than ten half-lives of the respective drug before enrolment in the study
* Use of any drugs, which might influence the results of the trial within two weeks prior to administration or during the trial
* Participation in another trial with an investigational drug (<= two months prior to administration or during trial)
* Smoker (> 10 cigarettes or > 3 cigars or > 3 pipes/day)
* Inability to refrain from smoking on study days
* Alcohol abuse (> 60 g/day)
* Drug abuse
* Blood donation (>= 100 mL within four weeks prior to administration or during the trial)
* Excessive physical activities (within the last week before the study)
* Any laboratory value outside the reference range of clinical relevance

Ages: 21 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2002-04; Primary Completion 2002-06 (Actual)

PRIMARY OUTCOMES:
Number of subjects with adverse events | up to 12 days after drug administration
Number of subjects with clinically significant findings in vital signs | up to 12 days after drug administration
  blood pressure, pulse rate, respiratory rate, oral body temperature
Number of subjects with clinically significant findings in ECG | up to 12 days after drug administration
Number of subjects with clinically significant findings in laboratory tests | up to 12 days after drug administration

SECONDARY OUTCOMES:
Plasma concentration time profiles | up to 96 hours after drug administration
Maximum measured concentration of the analyte in plasma (Cmax) | up to 96 hours after drug administration
Time from dosing to the maximum concentration of the analyte in plasma (tmax) | up to 96 hours after drug administration
Area under the concentration-time curve of the analyte in plasma from time zero to a specified point in time (AUC0-t) | up to 96 hours after drug administration
Terminal half-life of the analyte in plasma (t1/2) | up to 96 hours after drug administration
Mean residence time of the analyte in the body (MRT) | up to 96 hours after drug administration
Total clearance of the analyte in plasma (CL) | up to 96 hours after drug administration
Apparent volume of distribution at steady state (Vss) | up to 96 hours after drug administration
Amount of drug excreted into urine (Ae) | up to 72 hours after drug administration